CLINICAL TRIAL: NCT06075706
Title: A Randomised, Open-label, Controlled, Multicentre, Phase 2 Trial of First-line Treatment With Mesenchymal Stromal Cells MC0518 Versus Best Available Therapy in Paediatric Participants With Steroid-refractory Acute Graft-versus-host Disease After Allogeneic Stem Cell Transplantation (BALDER Trial)
Brief Title: Trial of Efficacy and Safety of MC0518 Versus Best Available Therapy in Participants With Steroid-Refractory Acute Graft Versus Host Disease
Acronym: BALDER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC-MSC.2/aGvHD; 2023-503952-28-00 (Other: EU CT Number)
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Steroid-refractory Acute Graft-versus-host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MC0518 (Experimental): Participants will be treated with intravenous infusions of MC0518 at a dose of 1 to 2*10^6 cells per kilogram (cells/kg) (based on body weight at the Screening Visit). Infusions will be administered once a week for 4 weeks (Visit Day 1, 8, 15, and 22). Participants with partial response (PR) on Day 28 will have 2 additional MC0518 infusions administered on Day 29 and 36.
  Interventions: Biological: MC0518
- Best Available Therapy (BAT) (Active Comparator): Participants will receive one of the following systemic BATs based on the Investigator's decision: extracorporeal photopheresis (ECP), anti-thymocyte globulin (ATG), etanercept, infliximab or ruxolitinib (RUX).
  Interventions: Biological: BAT

INTERVENTIONS:
Biological: MC0518 — MC0518 will be intravenously infused immediately after thawing.
  Arms: MC0518
Biological: BAT — BAT including ECP, ATG, etanercept, infliximab or RUX will be administered based on Investigator's decision.
  Arms: Best Available Therapy (BAT)

SUMMARY:
The purpose of this trial is the comparative evaluation of overall response rate (ORR) in paediatric participants with steroid-refractory acute graft-versus-host disease (SR-aGvHD) at Visit Day 28 after treatment with MC0518 or first used best available therapy (BAT).

ELIGIBILITY:
Inclusion Criteria:

1. Participant had a previous allogeneic HSCT as indicated for non-malignant (including inborn errors of metabolism, primary immunodeficiencies, haemoglobinopathies, and bone marrow failure syndromes) or hematological malignant disease or neuroblastoma.
2. Participant has been clinically diagnosed with Grade II to IV aGvHD according to Harris et al. A biopsy of the involved organs with aGvHD is encouraged but not required.
3. Participant has experienced failure of previous first-line aGvHD treatment (that is, SR-aGvHD), defined as:

   * aGvHD progression within 3 to 5 days of therapy onset with >=2 milligram per kilogram per day (mg/kg/day) of prednisone equivalent or
   * failure to improve within 5 to 7 days of treatment initiation with >=2 mg/kg/day of prednisone equivalent or
   * incomplete response after greater than (>) 28 days of immunosuppressive treatment including at least 5 days with >=2 mg/kg/day of prednisone equivalent.
4. Male or female participant who is >=28 days and <18 years of age and has a minimum body weight of 3.2 kilograms (kg) at the Screening Visit.
5. Participant has an estimated life expectancy of >28 days.
6. Participant, if female and of childbearing potential, agrees to use a highly effective contraceptive measure starting at the Screening Visit and continuing throughout the entire trial period.
7. Participant, if a fertile male, agrees to sexual abstinence or to use a condom during sexual activity with their female partner of childbearing potential or pregnant partner. Additionally, if their partner is a woman of childbearing potential (WOCBP), then their partner must use an additional highly effective contraceptive method during sexual activity starting at the Screening Visit and continuing throughout the entire trial period.
8. A written informed consent of the participant's parent(s) / legal guardian(s) (and participant's assent, when applicable) has been obtained according to national regulations.

Exclusion Criteria:

1. Participant has overt relapse or progression or persistence of the underlying disease.
2. Participant has received the last HSCT for a solid tumor disease other than neuroblastoma.
3. Participant has graft-versus-host disease overlap syndrome.
4. Participant has received systemic first-line treatment for aGvHD other than steroids and a prophylaxis with other than calcineurin inhibitors, mammalian target of rapamycin (mTOR) inhibitors, anti-thymocyte globulin, mycophenolate mofetil, methotrexate, abatacept, or cyclophosphamide. Note: In vitro or in vivo graft manipulation to prevent graft-versus-host disease (example, T-cell depletion) during HSCT is permitted. Restart of initial prophylaxis with calcineurin inhibitors, mammalian target of rapamycin inhibitors, or mycophenolate mofetil after aGvHD onset is permitted.
5. Participant has received prior mesenchymal stromal cell (MSC) treatment, including MC0518/Obnitix®.
6. Participant has a known pregnancy (as confirmed by a positive pregnancy test result at the Screening Visit) and / or is breastfeeding.
7. Participant has a known hypersensitivity to MC0518 and / or its excipients (dimethyl sulfoxide, human serum albumin, isotonic sodium chloride solution).
8. Participant has a known hypersensitivity or any contraindication to the Investigator's choice BAT (extracorporeal photopheresis, anti thymocyte globulin, etanercept, infliximab, or ruxolitinib) and / or its excipients. For a list of excipients please refer to the respective Summary of Product Characteristics.
9. Participant has an underlying or current medical or psychiatric condition that, in the opinion of the Investigator, would interfere with the evaluation of the participant.
10. Participant has an uncontrolled infection (examples, sepsis or multi-organ failure) including significant bacterial, fungal, viral, or parasitic infection requiring treatment.
11. Participant has received treatment with any other investigational agent within 30 days or 5 half-lives (whichever is longer) before the Screening Visit.

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Overall Response (OR) | At Day 28
  OR is defined as complete response (CR) or partial response (PR) at Day 28 relative to acute graft-versus-host disease (aGvHD) status at baseline. CR is defined as resolution of aGvHD in all involved organs. PR is defined as improvement in 1 stage in at least 1 or more organs involved with aGvHD symptoms without progression in others.

SECONDARY OUTCOMES:
Number of Participants With Freedom From Treatment Failure (FFTF) Until 6 Months (Day 180) | Up to 6 months (Day 180)
  FFTF is defined as the time from the date of randomization to the date of the event. An event is defined as death, relapse or progression of the underlying disease, or addition or change to any further systemic immunosuppressive aGvHD therapy.
Overall Survival (OS) | Up to Month 24
  Overall survival is defined as the time from randomization to the date of death due to any cause.
Number of Participants With aGvHD Response | At Days 28, 60, 100 and 180
  aGvHD response will be categorized as OR (CR + PR), CR, PR, and NR. NR is defined as the absence of CR or PR.
Change From Baseline in aGvHD Grades | Baseline, Days 8, 15, 22, 28, 60, 100 and 180
  aGvHD grades: Grade 0- no organ involvement (that is, Stage 0 skin, Stage 0 liver, and Stage 0 gastrointestinal [GI]); Grade I-Stage 1 - 2 skin without liver/GI involvement; Grade II- Stage 3 skin and / or Stage 1 liver and / or Stage 1 GI; Grade III- Stage 2 - 3 liver and / or Stage 2 - 3 GI; Grade IV- Stage 4 skin and / or Stage 4 liver and/or Stage 4 GI.
Time to Response | From the date of the first treatment administration to the date of the first response (CR or PR) (up to 5 years)
  Time to response is defined as the time from the date of the first treatment administration to the date of response (CR or PR).
Duration of Response | Up to Month 24
  Duration is defined as the time from the date of the first OR (CR or PR) to the date of aGvHD assessed as NR compared to the baseline assessment, or the date of addition of or change to any further systemic aGvHD therapy (except changes in steroid treatment), in responders.
Number of Participants With Best Overall Response (OR) | Up to Day 28
  Best OR is defined as the achievement of an OR at any time point up to and including Day 28.
Cumulative Dose of Steroids for SR-aGvHD per Kilogram (kg) of Body Weight | From the date of the first treatment administration up to Day 28, Day 60, and Month 24
  The cumulative dose of steroids given for SR-aGvHD per kg of body weight from the date of the first treatment administration until Day 28, Day 60, and until Visit Month 24 will be analyzed.
Number of Participants With Chronic Graft-versus-host Disease (cGvHD) | From Day 60 up to Month 24
  Number of participants with cGvHD will be reported.
Time to Chronic Graft-versus-host Disease (cGvHD) | From Day 60 up to Month 24
  Time to cGvHD is defined as the time between the last day of hematopoietic stem cell transplantation (HSCT) to the first episode of cGvHD.
Number of Participants With Graft Failure (GF) | Baseline up to Month 24
  Number of participants with GF will be reported.
Number of Participants With Relapse or Progression in Participants With Underlying Malignant Disease | From randomization up to Month 24
  Number of participants with relapse or progression in participants with underlying malignant disease will be reported.
Time to Relapse or Progression in Participants With Underlying Malignant Disease | From randomization up to Month 24
  Time to relapse or progression is defined as the time from the date of randomization to the date of relapse or progression until Month 24.
Event-free Survival (EFS) | From the date of randomization to date of GF, relapse or progression of the underlying disease, or death due to any cause, whichever occurs first (up to Month 24)
  EFS is defined as the time from the date of randomization to the date of the event. An event is defined as GF, relapse or progression of the underlying disease, or death due to any cause.
Non-relapse Mortality (NRM) | From the date of randomization to the date of death without previous relapse or progression of the underlying disease (up to Month 24)
  NRM is defined as the time from the date of randomization to the date of the event. An event is defined as death without previous relapse or progression of the underlying disease.
Number of Participants With Adverse Events (AEs) | Up to Month 24
  An AE is defined as any untoward medical occurrence in a trial participant administered a trial treatment that does not necessarily have a causal relationship with this trial treatment.
Number of Participants With Adverse Reactions (ARs) by Severity | Up to Month 24
  An AR is defined as all noxious and unintended responses to a trial treatment related to any dose administered / procedure performed. Severity will be graded based on Common Terminology Criteria for Adverse Events (CTCAE) v5.0: Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe; Grade 4- Life-threatening consequences; urgent intervention indicated; Grade 4- Death related to the AE.
Change From Baseline in Performance Score Based on Karnofsky Scale | Baseline, Days 8, 15, 22, 28, 60 and 100
  The Karnofsky performance score (KPS), which is reported on an ordinal scale from 0 to 100, provides a rough measure of the participant's (recipient age greater than or equal to [>=] 16 years) well-being, including their ability to conduct activities of daily living and functional capacity. Higher score indicates normal, no complaints and no evidence of disease.
Change From Baseline in Performance Score Based on Lansky Scale | Baseline, Days 8, 15, 22, 28, 60 and 100
  A Lansky score (recipient age >=1 year and less than [<] 16 years) will be recorded pre-treatment and measured serially at regular intervals after treatment. The score is a standard performance score that measures overall function of the child with a scale range from 0 to 100. Higher score indicates full activeness.
Pediatric Quality of Life Inventory (PedsQL™) 4.0 Generic Core Scale Score | Baseline, Days 28, 60, 100 and 180
  The PedsQL Generic Core Scales instrument is a standardized, established, and validated questionnaire in pediatric populations that systematically assesses the participants' and parents' / legal guardians' perceptions of health-related quality of life (HRQoL). The Generic Core Scales module consists of 23 items measuring the core dimensions of health on physical, emotional, social, and school functioning that can be used for self- and proxy-reports in age groups ranging from 2 to 18 years (child self-report ages: 5 to 7, 8 to 12, 13 to 18; parent-proxy report ages: 2 to 4, 5 to 7, 8 to 12, 13 to 18). The scores of this questionnaire range from 0 to 100 , where higher scores indicate better HRQoL.
Change From Baseline in PedsQL™ Stem Cell Transplant Module Scale Score | Baseline, Days 28, 60, 100 and 180
  The PedsQL™ Stem Cell Transplant Module is a disease-specific module of the PedsQL™ for toddlers (2 to 4 years of age), young children (5 to 7 years of age), children (8 to 12 years of age), and adolescents (13 to 18 years of age) and was designed to measure the quality of life in participants undergoing stem cell transplantation. It consists of the following HRQoL domains: pain and hurt, fatigue / sleeping problems / weakness, nausea, worry / anxiety about disease / treatment, nutritional problems, neurocognitive problems, communication about disease / treatment, loneliness, physical functioning and additional somatic complaints (pruritus, skin inflammation, oral problems, eyes or breathing) including patients' and parents' assessment. The scores of this disease-specific module of the PedsQL™ range from 0 to 100, where higher scores indicate better HRQoL.

CONTACTS AND LOCATIONS:
Locations (36):
- France (11):
  - CHU de Bordeaux - Hopital des Enfants, Bordeaux
  - CHU Grenoble Alpes - Hopital Couple Enfant (HCE), La Tronche
  - Centre Hospitalier Universitaire de Lille CHU Lille - Hopital Jeanne de Flandre HJF, Lille
  - Institut d'Hematologie et d'Oncologie Pediatrique (IHOPe), Lyon
  - CHU de Marseille-Hopital de la Timone, Marseille
  - Centre Hospitalier Regional Universitaire (CHRU) Montpellier - hopital Arnaud de Villeneuve, Montpellier
  - CHU de Nantes - Hopital Mere Enfant, Nantes
  - Hopital Robert Debre, Paris
  - CHU de Rouen - Hopital Charles Nicolle, Rouen
  - CHRU de Strasbourg - Hopital de Hautepierre, Strasbourg
  - CHRU Nancy, Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (9):
  - Uniklinik RWTH Aachen, Klinik fur Kinder- und Jugendmedizin, Aachen
  - Universitaetsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe, Frankfurt
  - Universitaetsklinikum Freiburg - Zentrum fuer Kinder- und Jugendmedizin (ZKJ), Freiburg im Breisgau
  - Justus-Liebig-Universitaet Giessen, Giessen
  - Medizinische Hochschule Hannover MHH, Hanover
  - Department of Pediatrics, Jena University Hospital, Jena
  - Universitaetsklinikum Leipzig - Abteilung fuer Paediatrische Onkologie, Haematologie und Haemostaseologie, Leipzig
  - Universitaetsklinikum Muenster (UKM) - Klinik fuer Kinder- und Jugendmedizin - Paediatrische Haematologie und Onkologie, Münster
- Italy (5):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico S.Orsola Malpighi, Bologna
  - Pediatric Clinic Onco Hematology San Gerardo Hospital, Monza
  - U.O.C. Oncoematologia Pediatrica, Fondazione IRCCS Policlinico San Matteo, Pavia
  - Hematology and Cellular Therapy Ospedale Bambino Gesu, Rome
  - A.O.U. Citta della Salute e della Scienza di Torino Ospedale Infantile Regina Margherita, Turin
- Poland (3):
  - Department of Pediatric Hematology, Oncology and BMT, Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship
  - Dzieciecy Szpital Kliniczny im. A.Gebali w Lublinie, Lublin
  - Szpital Kliniczny im. Karola Jonschera UM, Poznan
- Spain (8):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitario Vall dHebron, Barcelona
  - Hospital Sant Joan de Deu Barcelona (HSJDB), Barcelona
  - Hospital NiÃ±o Jesus, Madrid
  - Hospital Infantil Universitario La Paz, Madrid
  - Instituto de Investigacion Biomedica de Malaga IBIMA - sede Hospital Regional Universitario de Malaga HRUM Hospital Carlos Haya, Málaga
  - Instituto Murciano de Investigacion Biosanitaria (IMIB) Virgen de la Arrixaca, Murcia
  - Hospital Universitari I politecnic La Fe Jose, Valencia